CLINICAL TRIAL: NCT06845839
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously Administered CAY001 in Healthy Volunteer Subjects
Brief Title: Study to Evaluate CAY001 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cayuga Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAY001-01; MT21006.078 (Other Grant/Funding Number: Combat Casualty Care); MTEC-21-06-MPAI-078 (Other Grant/Funding Number: MTEC)
Record Dates: First submitted 2024-11-08; First posted 2025-02-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: hemorrhage; polyphosphate; hemostatic drug; coagulation; clotting
MeSH Terms: conditions — Hemorrhage; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAY001 (Experimental)
  Interventions: Drug: CAY001
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CAY001 — Polyphosphate (PolyP) - silica nanoparticle (SNP) complex
  Arms: CAY001
Other: Placebo — Vehicle - aqueous solution
  Arms: Placebo

SUMMARY:
This is a Phase 1, first-in-human, randomized, double-blind, placebo-controlled, single ascending dose, sequential group study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of CAY001 when administered to healthy male and female subjects. Three dose levels will be evaluated with a total of approximately 24 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to provide written informed consent
2. The subject is male or female (based on gender assigned at birth), 18-50 years of age inclusive
3. The subject has a body mass index ≥ 18 and ≤ 30.0 kg/m2 and weighs at least 61 kg for males and females
4. The subject is in good general health per Investigator evaluation for age as determined by medical history, vital signs, physical examination findings, screening laboratory test results, and 12-lead ECG results.

   Specific inclusionary laboratory values prior to randomization require the following.
   * Aspartate transaminase (AST), alanine transaminase (ALT) < 1.5 x upper limit of normal (ULN)
   * Total serum bilirubin and alkaline phosphatase levels < 1.2 x ULN
   * White blood cell (WBC) count, platelet count, and hemoglobin level within the normal range; out of range values are allowed if per the Investigator they are not deemed clinically significant
   * PT/INR, partial thromboplastin time (PTT), and D-dimer level (age-adjusted) within the normal range
5. Negative drug and alcohol tests at Screening and check-in (Day -1) and willing to abstain from alcohol and recreational drug use from the screening visit until the EOS/ET Visit;
6. No use of any tobacco or nicotine-containing products within 3 months, negative cotinine test at Screening and check-in (Day -1), and willing to abstain from tobacco or nicotine use from the screening visit until the EOS/ET Visit;
7. Male and female (women of childbearing potential [WOCBP]) subjects of childbearing potential must agree to the double-barrier method (i.e. male condom and spermicide or diaphragm and spermicide) or abstinence and refrain from sperm/egg donation throughout the study starting with the first dose of study treatment and for at least 3 months after the last dose of study drug. Hormonal contraceptives and intrauterine devices [IUD] must be stopped at least 3 months prior to the first dose of study treatment and for at least 3 months after the last dose of study drug. ▪ Note: Non-WOCBP includes healthy postmenopausal women who have undergone surgical menopause (hysterectomy, oophorectomy) or have been naturally menopausal, with no menstrual cycle for at least 24 months prior to Day 1; In the case of females, a negative serum pregnancy test (SPT) at Screening and a negative urine pregnancy test at check-in on Day -1.
8. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study

Exclusion Criteria:

1. Any clinically significant acute or chronic medical condition that in the evaluating Investigator's opinion could interfere with the study
2. Any history of plastic surgery involving silicone, any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the study drug or any planned surgical procedure that will occur during the study and cannot be delayed (from screening through the Day 28 EOS/ET Visit);
3. Any clinically significant abnormal findings in physical examination, vital signs, laboratory assessments (other than those discussed in the inclusion criteria), and ECG parameters identified during screening or check-in that in the evaluating Investigator's opinion could interfere with the study. Note: abnormal test results may be repeated once for confirmation;
4. Any of the following vital signs occurring after 10 minutes of supine rest at screening or check-in: ▪ Systolic blood pressure >140 mm Hg ▪ Diastolic blood pressure >90 mmHg ▪ Heart rate <45 or >100 beats per minute
5. Any of the following ECG parameters at screening or check-in:

   * Prolonged Fridericia-corrected QT interval (QTcF) >450 msec for males and > 460 msec for females, shortened QTcF <340 msec, or pause >3 seconds;
   * Prolonged PR (PQ) interval >200 msec, intermittent second- or third-degree atrioventricular (AV) block or AV dissociation
   * Complete right or left bundle branch block (QRS > 120 msec); left ventricular hypertrophy
   * Family history of long QT syndrome or sudden cardiac death
6. Have a known hypersensitivity or allergy to CAY001 components polyP or SNP, or to any ingredients in medication(s) to be received in this study;
7. Any history of significant liver, spleen, or kidney conditions
8. Any history of arterial or venous thrombosis or hypercoagulable or thrombotic condition, including any of the following

   * History of transient ischemic attack, cardiovascular accident, stroke (ischemic or hemorrhagic), unstable angina, myocardial infarction, or peripheral arterial disease
   * History of deep venous thrombosis, pulmonary embolus, thrombophlebilitis or arterial thrombosis
   * History of known clotting disorders like factor V leiden syndrome, protein C or S deficiency, or antiphospholipid syndrome;
9. An increased risk of bleeding, including but not limited to the following:

   * Recent history (within 6 months preceding the first dose of study drug) of gastrointestinal (GI) bleeding that required unscheduled medical evaluation;
   * History of intracranial, intraocular, retroperitoneal, or spinal bleeding;
   * Recent major trauma (within 6 months preceding the first dose of the study drug)
   * History of hemorrhagic disorders, e.g. hemophilia, von Willebrand's disease, Hermansky-Pudlak syndrome
   * History of severe head trauma, intracranial hemorrhage, intracranial neoplasm, arteriovenous malformation, aneurysm, or proliferative retinopathy;
   * Subject reported history of blood in the stool
10. Use of any prescription, investigational or illicit drugs within 30 days (or 5 half-lives whichever is longer) prior to dosing;
11. Use of any over-the-counter (OTC) products, dietary supplements and herbal products (ie. St. John's Wort or fish oil) within 14 days of dosing through the Day 7 Safety Follow-up Visit;
12. Known active hepatitis B or C infection, human immunodeficiency virus (HIV) infection, or known other immune deficiency disease at screening;
13. Females who are pregnant, plan to become pregnant within 3 months of the last dose of study drug, or are breastfeeding a child;
14. History of or treatment for alcoholism or drug addiction within 1 year;
15. Receipt of blood transfusion, blood-derived products, or coagulation factors within 1 month prior to Day 1;
16. Prior exposure to CAY001;
17. An employee, family member, or student of the Sponsor, Investigator, or clinical site(s);
18. Unable to adhere to or understand the requirements of the protocol.
19. Consume caffeine containing food or beverages 48 hours prior to check in and during study confinement period.
20. Females who are actively menstruating on the day of dosing (Day 1).
21. Subject meets eligibility criteria, but study is filled.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of serious adverse events from Baseline through Day 28. | 28 days
Incidence and severity of treatment related adverse events from Baseline through Day 28 | 28 days
Changes in physical examination findings from Baseline through Day 28 | 28 days
  Physical examination includes general appearance, HEENT (head, eyes, ears, nose, throat), chest/lungs, heart, abdominal, neurological, extremities, skin, and palpable lymph nodes. Physical examination will be conducted at screening, at multiple timepoints during the study (symptom-directed).
Changes in electrocardiograms (ECGs) from Baseline through Day 28 | 28 days
  A standard 12-lead ECG will be performed after at least 10 minutes in the supine position. ECG data collected includes PR, QT interval, QRS duration, QTcF and heart rate.
Changes in systolic and diastolic blood pressure in mmHg from Baseline through Day 28 | 28 days
  Vital signs, including blood pressure will be collected with the subject supine and after resting for 10 minutes.
Changes in blood chemistry parameters (calcium, phosphorus, glucose, BUN, uric acid, bilirubin, creatinine and magnesium) in mg/dL, from Baseline through Day 28 | 28 days
Changes in hematology parameters (white blood cell, red blood cell, platelets) in x10E3/uL, from Baseline through Day 28 | 28 days
Changes in coagulation parameters (aPTT and PT) in seconds, from Baseline through Day 28 | 28 days
Changes in urinalysis from Baseline through Day 28 | 28 days
  Urinalysis evaluations are microscopic examination and specific gravity, pH, protein, glucose, ketones, blood, urobilinogen, bilirubin, nitrites and leucocyte values.
Changes in temperature in degrees Celsius from Baseline through Day 28 | 28 days
  Vital signs, including temperature, will be collected with the subject supine and after resting for 10 minutes.
Changes in pulse in beats per minute, from Baseline through Day 28 | 28 days
  Vital signs, including pulse, will be collected with the subject supine and after resting for 10 minutes.
Changes in respiratory rate in breaths per minute, from Baseline through Day 28 | 28 days
  Vital signs, including respiratory rate, will be collected with the subject supine and after resting for 10 minutes.
Changes in blood chemistry (total protein, albumin) in g/dL, from Baseline through Day 28 | 28 days
Changes in blood chemistry (alkaline phosphatase, AST, ALT, GGT ) in IU/dL, from Baseline through Day 28 | 28 days
Changes in blood chemistry (creatinine kinase, ) in U/L, from Baseline through Day 28 | 28 days
Changes in blood chemistry (potassium, sodium, chloride) in mmol/L, from Baseline through Day 28 | 28 days
Changes in hematology parameters (hemoglobin, MCHC) in g/dL, from Baseline through Day 28 | 28 days
Changes in hematocrit in % from Baseline through Day 28 | 28 days
Changes in hematology parameter, MCV, in fL from Baseline through Day 28 | 28 days
Changes in hematology parameter, MCH in pg from Baseline through Day 28 | 28 days
Changes in coagulation parameter, D-Dimer, in mg/L FEU, from Baseline through Day 28 | 28 days
Changes in coagulation parameter, INR, in NA, from Baseline through Day 28 | 28 days

SECONDARY OUTCOMES:
Change in calibrated automated thrombogram-thrombin generation assay (CAT-TGA) from Baseline through Day 28 | 28 days
  CAT-TGA is an ex vivo assay to determine the speed and amount of thrombin generated.
Determine the half-life (t½) (terminal) | Pre-dose through 24 hours post-dose
  Pharmacokinetic assay
Determine the time to maximum concentration (Tmax) | Pre-dose through 24 hours post-dose
Determine the maximum observed concentration (Cmax) | Pre-dose through 24 hours post-dose
Determine the area under the curve (AUC) | Pre-dose through 24 hours post-dose
Determine the AUC zero to infinity (AUC0-∞) | Pre-dose through 24 hours post-dose
Determine the AUC zero to last measurable concentration (AUC0-last) | Pre-dose through 24 hours post-dose
Determine the clearance (CL) | Pre-dose through 24 hours post-dose
Determine the volume of distribution at steady state (Vss) | Pre-dose through 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Charles Pollack, MD, Study Director — Cayuga Biotech, Inc.
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No